CLINICAL TRIAL: NCT04900168
Title: A Multi-center Observational Cohort Study of Management of Moderate Traumatic Brain Injury With or Without Intracranial Pressure Monitoring in Patients With Moderate Traumatic Brain Injury in China
Brief Title: Intracranial Pressure Monitoring in Moderate Traumatic Brain Injury
Acronym: IPMMTBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202102-18
Record Dates: First submitted 2021-04-07; First posted 2021-05-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Moderate Traumatic Brain Injury
Keywords: Intracranial Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- ICP monitoring group: patients received ICP monitoring
  Interventions: Device: Intracranial pressure monitoring
- conventional treatment group: patients without ICP monitoring and received conventional treatment

INTERVENTIONS:
Device: Intracranial pressure monitoring — An invasive method to monitor the intracranial pressure of patient
  Groups: ICP monitoring group

SUMMARY:
Objectives The primary focus for scientific investigation is to conduct a multi-center observational study to determine if intracranial pressure (ICP) monitoring to direct treatment of patients with moderate traumatic brain injury (TBI) improves medical practice and patient outcomes in China.

Design and Outcomes This is a prospective observational cohort multi-center study with blinded evaluation of outcome. It is a 2-group design. Neurologic outcome is evaluated by extended Glasgow outcome score(GOSE) at 6 months.

Interventions and Duration This is an observational study. The decision of intracranial pressure monitoring is made by the relatives of patient. Management of all patients will be consistent with protocols presently being used in the study hospitals. For patients who received ICP monitoring, the management will also be based specifically on the presence of intracranial hypertension. Each patient will be evaluated at 6 months post injury on neurological outcomes.

Sample Size and Population 832 patients with moderate traumatic brain injury will be collected on this study.

ELIGIBILITY:
Inclusion Criteria:

* History of head trauma
* 18 ≤ age ≤ 70 years
* Abnormal head CT scan (skull fracture, intracranial hematoma, brain contusion, cerebral infarction, brain edema, hydrocephalus, etc.)
* Glasgow coma scale at admission: 9-12
* Arriving at hospital within 24 hours after injury
* Systolic blood pressure ≥100 millimeter of mercury
* No pregnant

Exclusion Criteria:

* Refusing follow up visit
* Penetrating head injury, spine or spinal cord injury
* Surgical treatment in other hospital before admission
* Cardiopulmonary resuscitation after injury or in need of blood transfusion due to active bleeding
* Consciousness disorder caused not by head trauma (alcoholism, drug overdose, etc.)
* Prior history of head trauma or stroke
* Multiple injuries, with severity score of other parts>18
* Rhabdomyolysis, with blood creatine kinase (CK)>5000 international unit/L
* Injury of aorta, carotid artery or vertebral artery
* Serum creatinine (female)>1.2mg/dL (106μmol/L), serum creatinine (male)>1.5mg/dL (133μmol/L)
* Glomerular filtration rate (eGFR) <60 milliliter/min
* Body mass index (BMI) <18.5kg/m2 or >40kg/m2
* Estimated survival time less than 1 year
* Participating in other on-going clinical researches
* Other systemic diseases: uremia, liver cirrhosis, malignant tumor, mental illness, drug, or alcohol dependence, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with acute moderate traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 832 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Good neurologic outcome | Within 6 months after traumatic brain injury
  The proportion of patients with good neurological outcomes (GOSE: 5-8) in each group at 6 months after traumatic brain injury

SECONDARY OUTCOMES:
6 months mortality | Within 6 months after traumatic brain injury
  The mortality of patients in each group at 6 months after traumatic brain injury
In-hospital mortality | Within 1 month after traumatic brain injury
  The mortality of patients in each group during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shannxi Province, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Godoy DA, Rubiano A, Rabinstein AA, Bullock R, Sahuquillo J. Moderate Traumatic Brain Injury: The Grey Zone of Neurotrauma. Neurocrit Care. 2016 Oct;25(2):306-19. doi: 10.1007/s12028-016-0253-y. PMID 26927279
- [Background] Hawryluk GW, Manley GT. Classification of traumatic brain injury: past, present, and future. Handb Clin Neurol. 2015;127:15-21. doi: 10.1016/B978-0-444-52892-6.00002-7. PMID 25702207
- [Background] Stocchetti N, Carbonara M, Citerio G, Ercole A, Skrifvars MB, Smielewski P, Zoerle T, Menon DK. Severe traumatic brain injury: targeted management in the intensive care unit. Lancet Neurol. 2017 Jun;16(6):452-464. doi: 10.1016/S1474-4422(17)30118-7. PMID 28504109
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Watanitanon A, Lyons VH, Lele AV, Krishnamoorthy V, Chaikittisilpa N, Chandee T, Vavilala MS. Clinical Epidemiology of Adults With Moderate Traumatic Brain Injury. Crit Care Med. 2018 May;46(5):781-787. doi: 10.1097/CCM.0000000000002991. PMID 29369057
- [Background] Lobato RD, Rivas JJ, Gomez PA, Castaneda M, Canizal JM, Sarabia R, Cabrera A, Munoz MJ. Head-injured patients who talk and deteriorate into coma. Analysis of 211 cases studied with computerized tomography. J Neurosurg. 1991 Aug;75(2):256-61. doi: 10.3171/jns.1991.75.2.0256. PMID 2072163
- [Background] Peterson EC, Chesnut RM. Talk and die revisited: bifrontal contusions and late deterioration. J Trauma. 2011 Dec;71(6):1588-92. doi: 10.1097/TA.0b013e31822b791d. PMID 22182868
- [Background] Compagnone C, d'Avella D, Servadei F, Angileri FF, Brambilla G, Conti C, Cristofori L, Delfini R, Denaro L, Ducati A, Gaini SM, Stefini R, Tomei G, Tagliaferri F, Trincia G, Tomasello F. Patients with moderate head injury: a prospective multicenter study of 315 patients. Neurosurgery. 2009 Apr;64(4):690-6; discussion 696-7. doi: 10.1227/01.NEU.0000340796.18738.F7. PMID 19197220
- [Background] Balestreri M, Czosnyka M, Hutchinson P, Steiner LA, Hiler M, Smielewski P, Pickard JD. Impact of intracranial pressure and cerebral perfusion pressure on severe disability and mortality after head injury. Neurocrit Care. 2006;4(1):8-13. doi: 10.1385/NCC:4:1:008. PMID 16498188
- [Background] Juul N, Morris GF, Marshall SB, Marshall LF. Intracranial hypertension and cerebral perfusion pressure: influence on neurological deterioration and outcome in severe head injury. The Executive Committee of the International Selfotel Trial. J Neurosurg. 2000 Jan;92(1):1-6. doi: 10.3171/jns.2000.92.1.0001. PMID 10616075
- [Background] Harary M, Dolmans RGF, Gormley WB. Intracranial Pressure Monitoring-Review and Avenues for Development. Sensors (Basel). 2018 Feb 5;18(2):465. doi: 10.3390/s18020465. PMID 29401746
- [Background] Steiner LA, Andrews PJ. Monitoring the injured brain: ICP and CBF. Br J Anaesth. 2006 Jul;97(1):26-38. doi: 10.1093/bja/ael110. Epub 2006 May 12. PMID 16698860
- [Background] Leinonen V, Vanninen R, Rauramaa T. Raised intracranial pressure and brain edema. Handb Clin Neurol. 2017;145:25-37. doi: 10.1016/B978-0-12-802395-2.00004-3. PMID 28987174
- [Background] Muballe KD, Sewani-Rusike CR, Longo-Mbenza B, Iputo J. Predictors of recovery in moderate to severe traumatic brain injury. J Neurosurg. 2018 Nov 9;131(5):1648-1657. doi: 10.3171/2018.4.JNS172185. Print 2019 Nov 1. PMID 30497133
- [Background] Li Z, Xu F, Li Y, Wang R, Zhang Z, Qu Y. Assessment of intracranial pressure monitoring in patients with moderate traumatic brain injury: A retrospective cohort study. Clin Neurol Neurosurg. 2020 Feb;189:105538. doi: 10.1016/j.clineuro.2019.105538. Epub 2019 Oct 31. PMID 31846845